CLINICAL TRIAL: NCT05636644
Title: Neoadjuvant Effect of Albumin Binding Paclitaxel Compared With Common Paclitaxel in Breast Cancer：an Observational Single Center Study of Clinical Efficacy in Adjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mei Zhang (Other)
Responsible Party: Sponsor-Investigator, Mei Zhang, Deputy chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXH2022ZX02167
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Paclitaxel，Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: anthracyclines+cyclophosphamide+other paclitaxel drugs
- Group B: anthracyclines+cyclophosphamide+nab paclitaxel
  Interventions: Drug: Taxol

INTERVENTIONS:
Drug: Taxol — All patients received TAC regimen: both groups received AC (epirubicin 75 mg/m ² and cyclophosphamide 500mg/m ²)， Group A was treated with docetaxel for 6 cycles every 3 weeks (75 mg/m on the first day ²)； Group B received six cycles of nab paclitaxel (125 mg/m ²)， every 3 weeks is a course of treatment.
  Groups: Group B

SUMMARY:
In recent years, the incidence rate of breast cancer has remained high. In China, breast cancer is the malignant tumor with the highest incidence rate among women. Although the research and development of various targeted drugs and the improvement of clinical treatment system have effectively improved the 5-year survival rate of breast cancer patients in China, the clinical treatment effect of breast cancer is still unsatisfactory. It is speculated that the main reasons for the poor clinical efficacy of breast cancer are drug tolerance, recurrence, distant metastasis, etc., which further leads to some limitations in the exploration of clinical drug development and regulatory mechanism. Paclitaxels are common chemotherapeutic drugs, which have been widely used in the treatment of breast cancer, ovarian cancer and some lung cancer. In2005, albumin binding paclitaxel was approved by FDA for the treatment of breast cancer patients. It is highly hydrophobic and requires a mixture of polyethylene castor oil and ethanol. These solvents will increase the toxic reactions of patients treated with paclitaxel, including severe allergic and anaphylactic reactions, and irreversible peripheral neuropathy, usually requiring the use of corticosteroids and antihistamines in advance.In order to further confirm the advantages of albumin binding paclitaxel and common paclitaxel chemotherapeutic drugs in neoadjuvant chemotherapy of breast cancer, this project intends to explore albumin binding based on different molecular types of breast cancer (luminal a, B, HER2 +, triple negative) An observational study on the efficacy of neoadjuvant chemotherapy with a-paclitaxel and common paclitaxel chemotherapeutic drugs. Randomized grouping confirmed the effectiveness of albumin binding paclitaxel replacing common paclitaxel in neoadjuvant chemotherapy of breast cancer with different molecular types, providing evidence-based medical evidence for the selection of paclitaxel chemotherapeutic drugs based on breast cancer molecular types. At the same time, the patients with poor efficacy among the patients who selected the neoadjuvant chemotherapy scheme for breast cancer according to the guidelines of NCCN and CSCO were screened for clinical transformation research (including basic experimental research, follow-up intensive treatment selection, and providing basis for entering other drug clinical trials). For the patients who achieved the clinical efficacy of PCR with neoadjuvant chemotherapy, we further analyzed the reasons to explore a better scheme of neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female breast cancer patients aged ≥ 20 years and ≤ 70 years, with informed consent and meeting the treatment standard of neoadjuvant chemotherapy scheme; 2. Invasive breast cancer with TNM stageT2-4N0-3M0; 3.No treatment for breast cancer before enrollment, such as chemotherapy, targeted therapy and endocrine therapy; 4.All patients underwent thick needle biopsy of breast tumors (patients suspected of axillary lymph node metastasis should undergo lymph node biopsy) to determine the status of ER, PR, HER-2 and Ki-67; 5. All patients had normal cardiopulmonary function, liver and kidney function.

Exclusion Criteria:

* 1. The patient does not cooperate and is unwilling to sign the informed consent form; 2. The tumor has been confirmed to have distant metastasis; 3. Antitumor therapy, hormone replacement therapy and other breast cancer related treatments were performed before enrollment; 4. Any other malignant tumor is combined; 5. Patients with active infection, HIV history or chronic hepatitis B or C; 6. Persons with abnormal heart and lung functions or liver and kidney functions; 7.Other clinical researchers in recent 3 months.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with TNM stage T2-4N0-3M0 who were hospitalized in the breast surgery department of Shandong Qianfoshan Hospital from the time when the ethical approval document was obtained to December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission (pCR) | June 2025
  Grade I: tumor focus basically unchanged; Grade II: ≤ 30% tumor cells disappear; Grade III: about 30-90% of tumor tissues disappear; Grade IV: ≥ 90% of tumor cells disappeared; Grade V: no residual invasive cancer tissue. Among them, if there is grade III or above, it indicates that the treatment is effective; if there is grade II or below, it indicates that the treatment is invalid; and grade V 5 indicates that the patient has reached pCR.

SECONDARY OUTCOMES:
Disease free survival (DFS) | June 2025
Complete remission (CR), partial remission (PR) and objective remission rate (ORR) of solid tumors | June 2025
  ① Complete remission (CR): all cancer foci disappeared, no new tumor foci appeared and maintained for at least 4 weeks; ② Partial remission (PR): the sum of the maximum diameters of tumor lesions decreased by ≥ 30% for at least 4 weeks; ③ Disease stability (SD): the sum of the largest diameters of tumor lesions decreased to PR, or increased to PD; ④ Disease progression (PD): The sum of the maximum diameters of tumor lesions increases by at least 20%, and its absolute value increases by at least 5 mm. The appearance of new lesions is also called PD. If the tumor has CR and PR, the original scheme is proved to be effective, and continue to treat according to the original scheme; In case of PD and SD, replace the scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Guoming Liu, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital); Yonghao Li, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital); Xinlei Zhang, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital); Ximei Sun, master, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital)
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided